CLINICAL TRIAL: NCT01837823
Title: YELLOW II Study: Reduction in Coronary Yellow Plaque, Lipids and Vascular Inflammation by Aggressive Lipid Lowering
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Texas Heart Institute (Wafic Said Molecular Cardiology Research Lab) (Unknown); AstraZeneca (Industry); InfraReDx (indirect) (Unknown)
Responsible Party: Principal Investigator, Annapoorna Kini, Professor of Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 12-1507; HS#: 12-00741
Record Dates: First submitted 2013-04-05; First posted 2013-04-23 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Obstructive Coronary Artery Disease; Coronary Artery Disease
Keywords: Coronary artery disease; Lipid; Regression; Plaque
MeSH Terms: conditions — Coronary Artery Disease; Plaque, Amyloid | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rosuvastatin (Experimental): All subjects will receive rosuvastatin 40mg/day
  Interventions: Drug: rosuvastatin

INTERVENTIONS:
Drug: rosuvastatin — All subjects will receive rosuvastatin 40mg/day for 8-12 weeks
  Other Names: Crestor

SUMMARY:
Coronary artery disease (CAD) remains a leading cause of death in most countries. It is well known that the reduction of cholesterol levels by statin therapy is associated with significant decreases in plaque burden. REVERSAL, ASTEROID, and more recently the SATURN II trial showed that in patients with CAD, lipid lowering with atorvastatin or rosuvastatin respectively reduced progression of coronary atherosclerosis, even causing plaque regression of some lesions. CAD clinical events are related to plaque instability due to lipid content and activity within the atherosclerotic plaque. The investigators recently completed the YELLOW I study, and identified that intensive statin therapy (rosuvastatin 40mg) was associated with a reduction in the amount of lipid in obstructive coronary plaques, as measured by near-infrared spectroscopy (NIRS). The YELLOW II study is designed to expand and build upon these results, and to provide mechanistic insights into the potential benefits of intensive statin therapy on atherosclerotic plaques.

DETAILED DESCRIPTION:
YELLOW II is a single site study and will assess the regression of plaque lipid content and changes in plaque morphology from atherosclerotic lesions after high-dose statin therapy by utilizing NIRS, IVUS and optical coherency tomography (OCT) imaging modalities in the coronary arteries. We propose to image non-culprit coronary lesions using these modalities in patients with two or three diseased coronary vessels deemed to warrant intervention on clinical grounds. Thus, at the time of enrolment patients will undergo Percutaneous Coronary Intervention (PCI) of a non-study culprit lesion, and triple-modality imaging of the potential non-culprit ('YELLOW') lesion. If there is high baseline lipid content in the non-culprit YELLOW lesion (max 4mm LCBI > 150), patients will be formally entered into this study. Following this, all enrolled subjects will receive high-dose lipid lowering therapy (rosuvastatin 40mg daily). The non-culprit YELLOW lesion will undergo staged intervention 8-12 weeks following study enrolment and baseline imaging. At this time the YELLOW lesion will be reimaged to determine whether high-dose statin therapy caused a reduction in lipid content as assessed by NIRS, and other altered plaque morphology as assessed by OCT and IVUS. In addition, both at baseline and at the time of final non-culprit YELLOW lesion PCI, blood samples will be drawn during baseline and follow-up procedure to characterize reverse cholesterol transport by ability of patient HDL to accept cholesterol from cholesterol-laden (mouse J774) macrophage (cholesterol efflux) and the effect of patient HDL and apolipoprotein A1 on macrophage gene expression and migration.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age and willing to participate.
* Fluency in either English or Spanish.
* Stable patients who will undergo cardiac catheterization and PCI (intent to stent).
* Patient is willing to go on high-dose cholesterol lowering medication for the duration of the study
* Signed written Informed Consent.
* Women of childbearing potential must agree to be on an acceptable method of birth control/contraceptive such as barrier method (condoms/diaphragm); hormonal contraceptives (birth control pills, implants (Norplant) or injections (Depo-Provera)); Intrauterine Device.
* Proposed non-culprit YELLOW study lesion with max 4mm LCBI ≥ 150.

Exclusion Criteria:

* Patients who have acute myocardial infarction (ST-segment elevation presentation, new Q waves or non-ST segment elevation with CK-MB > 5 times above the upper normal (31.5 ng/ml) within 72 hours).
* Patients who are in cardiogenic shock.
* Patients requiring coronary artery bypass graft surgery.
* Patients with platelet count < 100,000 cell/mm3.
* Patients who have co-morbidity which reduces life expectancy to one year.
* Patients who are currently participating in another investigational drug/device study.
* Patients with liver disease.
* Patient with creatinine > 2.0 mg/dL.
* Pregnant women and women of childbearing potential who intend to have children during the duration of the trial.
* Patients having undergone heart transplantation, or those that may undergo heart transplantation during the study period.
* Active autoimmune disease.
* Nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2013-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annapoorna Kini, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Jason Kovacic, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Kini AS, Vengrenyuk Y, Shameer K, Maehara A, Purushothaman M, Yoshimura T, Matsumura M, Aquino M, Haider N, Johnson KW, Readhead B, Kidd BA, Feig JE, Krishnan P, Sweeny J, Milind M, Moreno P, Mehran R, Kovacic JC, Baber U, Dudley JT, Narula J, Sharma S. Intracoronary Imaging, Cholesterol Efflux, and Transcriptomes After Intensive Statin Treatment: The YELLOW II Study. J Am Coll Cardiol. 2017 Feb 14;69(6):628-640. doi: 10.1016/j.jacc.2016.10.029. Epub 2016 Oct 29. PMID 27989886

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in July 2013, with enrollment from August 2013 to February 2015, 91 patients with multivessel CAD, who underwent percutaneous coronary intervention (PCI) for a culprit lesion followed by OCT and NIRS/IVUS imaging of an obstructive NCL were enrolled.
Groups:
- Rosuvastatin: All subjects will receive rosuvastatin 40mg/day 8-12 weeks
Period: Overall Study
Arm/Group | Rosuvastatin
Started | 91
Completed | 85
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 27
Hypertension [Count of Participants; unit: Participants] | 76
Hypercholesterolemia [Count of Participants; unit: Participants] | 75
Diabetes mellitus [Count of Participants; unit: Participants] | 37
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.6 (5.2)
Current smoking [Count of Participants; unit: Participants] | 12
History of smoking [Count of Participants; unit: Participants] | 26
Prior myocardial infarction (MI) [Count of Participants; unit: Participants] | 12
Prior percutaneous coronary intervention (PCI) [Count of Participants; unit: Participants] | 24
Statin use [Count of Participants; unit: Participants]
  atorvastatin | 29
  simvastatin | 23
  rosuvastatin | 12
  pravastatin | 4
  fluvastatin | 1
  none | 16
Location of coronary artery disease [Count of Participants; unit: Participants]
  the left anterior descending artery (LAD) | 36
  left circumflex artery (LCX) | 23
  the right coronary artery (RCA) | 26

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Plaque Morphology and HDL Functionality
Description: Correlation between the changes in plaque morphology composition by intravascular imaging with changes in HDL functionality. HDL functionality is measured by the Cholesterol Efflux Capacity (CEC). Plaque morphology is represented by the Fibrous Cap Thickness.
Time Frame: baseline and 8-12 weeks
Measure: Number (95% Confidence Interval); unit: beta coefficient
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 85
beta coefficient | 0.30 [0.07 to 0.54]

2. Primary Outcome: Correlation Between the Change in Fibrous Cap Thickness and Hs-CRP
Description: Correlation between the change in plaque morphology composition by intravascular imaging with inflammatory cell activity.
Time Frame: baseline and 8-12 weeks
Measure: Number (95% Confidence Interval); unit: beta coefficient
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 85
beta coefficient | -0.27 [-0.46 to -0.02]

3. Secondary Outcome: Maximal 4mm Lipid Core Burden Index (LCBI 4mm Max)
Description: Maximum LCBI 4mm (ΔLCBI4mm max) of the non-culprit YELLOW lesion at baseline and 8-12 weeks thereafter.
  LCBI4mm max : 4-mm long segment with maximum lipid core burden index (LCBI), where the LCBI is calculated as the fraction of yellow pixels on a chemogram x 1000. Each pixel on the chemogram represents a probability of lipid presence in the given region; pixels are color-coded on a red-to-yellow color scale, with the low probability of lipid shown as red and the high probability of lipid shown as yellow.
Time Frame: baseline and at 8-12 weeks
Measure: Mean (Standard Deviation); unit: LCBI4mm max
Groups:
- Baseline: Prior to rosuvastatin therapy
- 8-12 Weeks: After 8-12 weeks of rosuvastatin
Arm/Group | Baseline | 8-12 Weeks
Number analyzed (Participants) | 85 | 85
LCBI4mm max | 416.6 (172.9) | 400.2 (180.4)

4. Secondary Outcome: Fibrous Cap Thickness (FCT) by OCT
Description: ΔFibrous Cap Thickness measured by OCT at baseline and at 8-12 weeks
Time Frame: baseline and at 8-12 weeks
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Baseline | 8-12 Weeks
Number analyzed (Participants) | 85 | 85
μm | 100.9 (41.7) | 108.6 (39.6)
Statistical Analysis 1: Comparison: Baseline vs 8-12 Weeks; Test type: Superiority or Other; p = 0.054, Regression, Linear; Pearson correlation coefficient = -0.231

5. Secondary Outcome: IVUS Imaging Measures
Description: Correlation between ΔLCBI4mm max will be related to Δ values from baseline to 8-12 weeks thereafter in specific IVUS (ΔPlaque burden) imaging measures. Plaque burden is Plaque + Media divided by Total Plaque Area in %.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: percent of plaque burden
Arm/Group | Baseline | 8-12 Weeks
Number analyzed (Participants) | 85 | 85
percent of plaque burden
  Reference Site | 38.75 (10.54) | 38.93 (10.57)
  Minimum Lumen Area Site | 75.93 (7.07) | 75.79 (7.96)
Statistical Analysis 1: Comparison: Baseline vs 8-12 Weeks; for minimum lumen area site; Test type: Superiority or Other; p = 0.50, Pearson correlation coefficient; Pearson correlation coefficient = 0.074

6. Secondary Outcome: Inflammatory and Lipid Parameters
Description: ΔLCBI4mm max will be related to Δ values from baseline to 8-12 weeks thereafter in inflammatory and lipid parameters responses to patient-derived samples.
Time Frame: baseline and at 8-12 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Baseline | 8-12 Weeks
Number analyzed (Participants) | 85 | 85
mg/dl
  Total Cholesterol | 153.3 (44.9) | 115.0 (29.9)
  LDL Cholesterol | 86.8 (39.6) | 50.6 (25.0)
  HDL Cholesterol | 41.2 (12.7) | 42.2 (13.1)
  Triglyceride | 128.6 (111.8) | 107.8 (66.7)
  ApoB | 79.6 (28.0) | 57.4 (17.5)
  Apo-AI | 120.1 (25.6) | 126.9 (23.3)
  hs-CRP | 35.0 (55.0) | 27.0 (42.0)

7. Secondary Outcome: Lesion LCBI
Description: As related to other outcomes, change in LCBI measured across the entire lesion (rather than ΔLCBI4mm max). The LCBI Score, computed as the fraction of valid pixels within the scanned region that exceeded a LCP probability of 0.6 multiplied by 1000, summarized the amount of LCP in the entire scanned region of the coronary vessel on a 0-to-1000 scale .
Time Frame: at baseline and at 8-12 weeks
Measure: Median (Inter-Quartile Range); unit: LCBI4mm max
Arm/Group | Baseline | 8-12 Weeks
Number analyzed (Participants) | 85 | 85
LCBI4mm max | 142.84 [88.74 to 215.80] | 141.93 [96.92 to 239.21]

8. Secondary Outcome: LCBI 4mm at Same Anatomical Site
Description: As related to other outcomes, change in LCBI 4mm measured at the identical anatomical site at both time points, as defined by the LCBI4mm max site at baseline (rather than ΔLCBI4mm max).
  LCBI4mm: 4-mm long segment with maximum lipid core burden index (LCBI), where the LCBI is calculated as the fraction of yellow pixels on a chemogram x 1000. Each pixel on the chemogram represents a probability of lipid presence in the given region; pixels are color-coded on a red-to-yellow color scale, with the low probability of lipid shown as red and the high probability of lipid shown as yellow.
Time Frame: at baseline and at 8-12 weeks
Measure: Mean (Standard Deviation); unit: LCBI4mm max
Arm/Group | Baseline | 8-12 Weeks
Number analyzed (Participants) | 85 | 85
LCBI4mm max | 416.6 (172.9) | 383.2 (188.2)

9. Secondary Outcome: Change in Atheroma Volume
Description: Change in total atheroma volume (TAV) and lumen cross sectional area on OCT.
Time Frame: baseline and at 8-12 weeks
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Baseline | 8-12 Weeks
Number analyzed (Participants) | 85 | 85
mm^3 | 182.3 (94.5) | 182.7 (95.5)

10. Secondary Outcome: Biomarker Release
Description: Post procedure CK-MB, Troponin-I release at final YELLOW lesion PCI.
Time Frame: within 24 hrs of PCI
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 85
ng/ml
  CK-MB | 30. (3.5)
  Troponin-I | 0.35 (1.22)

11. Secondary Outcome: Correlation of Baseline Lipid Parameters With Baseline LCBI4mm Max
Description: Correlation of baseline lipid parameters with baseline LCBI4mm max
Time Frame: baseline
Measure: Number (95% Confidence Interval); unit: Beta coefficient
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 85
Beta coefficient | 0.07 [-0.64 to 1.27]

12. Secondary Outcome: Plaque Morphology as Related to Haptoglobin
Description: To relate changes in plaque lipid content and morphology to the patient haptoglobin genotype.
Time Frame: baseline and at 8-12 weeks
Population: Only those participants with these genotypes were analyzed
Measure: Mean (Standard Deviation); unit: LCBI4mm max
Groups:
- Hp2-2: Hp2-2 genotype
- Hp1-1/Hp 1-2: Hp1-1 or Hp 102 genotype
Arm/Group | Hp2-2 | Hp1-1/Hp 1-2
Number analyzed (Participants) | 31 | 54
LCBI4mm max
  Baseline | 440.3 (171.8) | 403.0 (173.7)
  at 8-12 weeks | 411.0 (201.5) | 393.9 (168.8)

13. Secondary Outcome: Mechanism of Reverse Cholesterol Transport
Description: To assess the mechanism of reverse cholesterol transport that arises with high-dose statin therapy, as related to changes in plaque lipid content and morphology, and systemic vascular inflammation. Reverse cholesterol transport (RCT) is a pathway by which accumulated cholesterol is transported from the vessel wall to the liver for excretion, thus preventing atherosclerosis.
Time Frame: baseline and at 8-12 weeks
Measure: Mean (Standard Deviation); unit: percentage of cholesterol
Arm/Group | Baseline | 8-12 Weeks
Number analyzed (Participants) | 85 | 85
percentage of cholesterol | 0.81 (0.14) | 0.84 (0.14)

14. Secondary Outcome: Correlation of Changes in Plaque Morphology
Description: Correlation of changes in plaque morphology by OCT, IVUS and NIRS with the perturbations in peripheral blood mononuclear cell transcriptome using microarray analysis.
  data not collected for this measure.
Time Frame: baseline and at 8-12 weeks
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 0

15. Secondary Outcome: MACE
Description: Major Adverse Cardiac Events (MACE) defined as a combined clinical endpoint of death, MI (Q wave or non Q-wave with CK-MB >3 times above the upper normal limit (48 U/L), urgent revascularization or stroke at 30 days.
Time Frame: at 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 85
Participants
  Myocardial infarction | 1
  Revascularization | 2
  Stroke | 0

16. Secondary Outcome: MACE
Description: Major Adverse Cardiac Events (MACE) defined as a combined clinical endpoint of death, MI (Q wave or non Q-wave with CK-MB >3 times above the upper normal limit (48 U/L), urgent revascularization or stroke at 1 year.
Time Frame: at 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 85
Participants | 33

ADVERSE EVENTS:
Arm/Group | Rosuvastatin
Serious Adverse Events (participants affected / at risk) | 3/85
Other Adverse Events (participants affected / at risk) | 30/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin (N=85)
Myocardial infarction (Cardiac disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin (N=85)
Urgent revascularization (Vascular disorders) | 13 (13)
Periprocedural complication (Surgical and medical procedures) | 2 (2)
Hospitalization for chest pain (Cardiac disorders) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes